CLINICAL TRIAL: NCT02214927
Title: Relative Bioavailability of 10 mg BI 11634 Immediate Release Tablet (IR) Compared to 10 mg of Oral Solution Following Oral Administration in Healthy Male Volunteers (Open-label, Single-dose, Intra-individual Comparison); Determination of Pharmacokinetics of 5 mg, 10 mg and 25 mg IR-tablet Formulation (Open-label, Single Dose)
Brief Title: Pharmacokinetics and Relative Bioavailability of 11634 Immediate Release Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1234.12
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — N-(1-(5-chloro-1H-benzimidazol-2-yl)-2-methoxyethyl)-3-methyl-4-(3-oxo-4-morpholinyl)benzamide

ARMS (2):
- BI 11634 single rising dose (Experimental): tablet
  Interventions: Drug: BI 11634 tablet
- BI 11634 cross-over (Experimental): sequence: 1. tablet 2. drinking solution
  Interventions: Drug: BI 11634 tablet; Drug: BI 11634 drinking solution

INTERVENTIONS:
Drug: BI 11634 tablet
Drug: BI 11634 drinking solution
  Arms: BI 11634 cross-over

SUMMARY:
* Characterisation of the relative bioavailability of the IR-tablet vs. oral drinking solution (no primary endpoint in a statistical sense)
* Safety and tolerability of the IR-tablet formulation and solution
* PK profile of the single ascending doses of the IR-tablet formulation (including analysis of dose proportionality)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian males according to the following criteria, based upon a complete medical history, including the physical examination, vital signs (blood pressure, pulse rate), 12-lead ECG, clinical laboratory tests
* Age ≥18 and ≤50 years
* Haemoglobin within the normal ranges
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Relevant surgery of gastrointestinal tract
* History of any bleeding disorder or acute and chronic blood coagulation defect, for the subject itself or any person of his family as far as known
* History of gastric ulcera and cholecystectomy
* Occult blood in faeces
* Relevant diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Relevant chronic or acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Use of acetylsalicylic acid or any other non-steroidal anti-inflammatory drugs (NSAID) within 2 weeks of study start until the end of study
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Alcohol abuse (more than 40 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Vulnerable subjects (e.g. persons kept in detention)
* Inability to understand and comply with protocol requirements, instructions and protocol-stated restrictions, the nature, scope and possible consequences of the study
* Subjects (including those who have had a vasectomy) who do not agree to use two methods of contraception, including barrier contraception (latex condoms with spermicide plus intrauterine device) when engaging in sexual activity with women of child bearing potential during the study and for 60 days after completion of the study
* Subjects with a history within the past six weeks of closed-head or torso trauma or deceleration injury such as an automobile accident or fall from a significant height

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 10 days after drug administration
Number of subjects with clinically significant findings in vital signs (blood pressure, pulse rate) | up to 10 days after drug administration
Number of subjects with clinically significant findings in ECG | up to 10 days after drug administration
Number of subjects with clinically significant findings in laboratory tests | up to 10 days after drug administration
Assessment of tolerability by investigator on a 4-point scale | up to 10 days after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration

SECONDARY OUTCOMES:
tmax (time from dosing to maximum measured concentration) | up to 24 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 up to the last quantifiable data point) | up to 24 hours after drug administration
λz (terminal rate constant in plasma) | up to 24 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 24 hours after drug administration
CL/F (apparent clearance of the analyte in plasma after extravascular administration) | up to 24 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 24 hours after drug administration
Activated partial thromboplastin time (aPTT) ratios between groups | up to 24 hours after drug administration
Maximum aPTT prolongation | up to 24 hours after drug administration
% inhibition of endogenous Factor Xa | up to 24 hours after drug administration
  by Russel's Viper Venom test (RVV)
Maximum international normalized ratio (INR) | up to 24 hours after drug administration
  compared between groups
Percent inhibition of thrombin generation by BI 11634 | up to 24 hours after drug administration
Percent peak inhibition of thrombin generation | up to 24 hours after drug administration
Time to maximum inhibition of thrombin generation BI 11634 | up to 24 hours after drug administration
Percent prolongation of lag time | up to 24 hours after drug administration
Area under the inhibition of the endogenous thrombin generation-time curve | up to 24 hours after drug administration
Maximum prolongation of blood coagulation time | up to 24 hours after drug administration
  by HepTest® (Haemachem Inc.) and COAMATIC® Heparin test (Chromogenix)
t1/2 (terminal half-life of the analyte in plasma) | up to 24 hours after drug administration